CLINICAL TRIAL: NCT03379272
Title: CONNECT: Comparison Of NeuroNaute Smart System to a Standard EleCTroencephalogram System in Hospital
Brief Title: Comparison Of NeuroNaute Smart System to a Standard EleCTroencephalogram System in Hospital
Acronym: CONNECT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Device evolves.
Sponsor: BioSerenity (Industry)
Collaborators: Pitié-Salpêtrière Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: n°2016-A01754-47
Record Dates: First submitted 2016-12-07; First posted 2017-12-20 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2020-12

CONDITIONS: Epilepsy
Keywords: Electroencephalography; Epilepsy; EEG
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GOLD STANDARD (Active Comparator): RECORDING WITH EEG GOLD STANDARD
  Interventions: Device: GOLDSTANDARD
- NEURONAUTE (Experimental): RECORDING WITH THE NEURONAUTE
  Interventions: Device: NEURONAUTE

INTERVENTIONS:
Device: GOLDSTANDARD — RECORDING WITH EEG GOLDSTANDARD
  Arms: GOLD STANDARD
Device: NEURONAUTE — RECORDING WITH NEURONAUTE
  Arms: NEURONAUTE

SUMMARY:
The proposed study is designed to evaluate the performance of the Neuronaute in comparison with the gold standard EEG in patients with a regular appointment at the hospital. The design of this study is guided by two overriding factors : (i) epileptics disorders suspected or either (ii) epileptics already diagnosed.

Volunteers will be asked to participate to this study. This study will enroll 35 outpatient subjects aged 18 to 85. Informed consent will be obtained from the patients, and assent from the subjects, prior to any form of assessment or intervention as part of the study.

Patients will be submitted to the studied device record Neuronaute following by the gold standard EEG.

A grid with all EEG activity recorded during the trial will be provided for evaluation after completion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients, with a regular appointment to perform an EEG recording: (i) suspected of epileptic disorders or (ii) epilepsy already diagnosed.
* Age (> 18 years),
* Affiliated to the social security
* Informed consent.

Exclusion Criteria:

* No informed consent
* Age (< 18 years)
* No affiliation to the social security
* Unsuitable anthropometric parameters
* Pregnant women
* Recent brain surgery
* Wound or scores on the body and the scalp
* Ongoing participation in another clinical trial
* Allergy to any component from MD including : Silver, polyamide, silicone
* Sensory disorders making the patient insensitive to pain on the skin
* Behavioral disorders making the patient excessively agitated or aggressive;
* Motor or mental disorders preventing the patient from expressing his or her pain;
* Cardiorespiratory disorders likely to be aggravated by slight compression of the chest;
* The susceptibility to tension headaches (the compression exerted by the bonnet may in certain cases trigger a headache)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-20 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of electroencephalographic signals interpretation recorded by the Neuronaute compared to the gold standard. | 1 year
  The main evaluation criteria is the reproducibility based on the interpretation of electroencephalographic signals recorded by the Neuronaute compared to the gold standard. The system will be considered effective if there are no significant differences in the physiological parameters recorded by the two systems.
  A clinical expert will interpret the EEG(electroencephalography) signals and fill the EEG evaluation sheet. It includes items such as signals quality and presence of abnormal events

SECONDARY OUTCOMES:
The Neuronaute will be considered effective if it detects inter-critical epileptic abnormalities in at least one patient. | 1 year
  A section of the evaluation sheet is designed for the secondary objectives.
The Neuronaute will be considered efficient if the installation time is at least as fast as the installation of the gold standard. The time will be measured from the beginning of the patient's preparation until the beginning of the recording. | 2 hours
  The time needed to set up the clinical device and the device under test will be noted in the Case Report Form.
The quality of the Neuronaute's ECG signal will be compared with the gold standard using an evaluation grid. | 1 year
  An evaluation grid led to compare the quality of th Neuronaute's ECG signal and Gold Standard' signal

IPD SHARING:
Plan to Share IPD: No